CLINICAL TRIAL: NCT06756217
Title: 68Ga-grazytracer PET/CT for Early Assessment of Response to Neoadjuvant Immunotherapy in Resectable NSCLC
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RTS-024
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3-5 tumor samples of typical cases will be collected for flow cytometric analysis and destroyed after test.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 68Ga-grazytracer PET/CT — 68Ga-grazytracer is designed to target granzyme B, and showed excellent in vivo metabolic stability and favorable targeting efficiency during immune responses. 68Ga-grazytracer PET/CT could directly display the killing effect of CD8+T cells on tumor. All enrolled patients underwent the same 68Ga-grazytracer PET/CT imaging.

SUMMARY:
The purpose of this study is to explore the effectiveness of 68Ga-grazytracer PET/CT in early evaluation of neoadjuvant immunotherapy response in resectable NSCLC.

DETAILED DESCRIPTION:
It is challenging to noninvasively early evaluate the immunotherapy response of cancer. The study will evaluate the application value of 68Ga-grazytracer PET/CT in the early evaluation of neoadjuvant immunotherapy response in resectable non-small cell lung cancer (NSCLC). Potential participants will be assessed for inclusion, including the verification of clinical stage and eligibility. Eligible patients with clinically stage IB-IIIA NSCLC will be received standardized neoadjuvant immunotherapy (every 3 weeks for 3 cycles). Patients with nonsquamous NSCLC will be received pembrolizumab plus platinum-pemetrexed, and lung squamous cell carcinoma patients will be received pembrolizumab plus platinum-paclitaxel. 68Ga-grazytracer PET/CT imaging will be performed at baseline and before cycle 3. Pathological response of the primary (MPR vs. Non-MPR), imaging response (iPR vs. Non-iPR; MR vs. MD), and 68Ga-grazytracer PET/CT imaging (Positive vs. Negative) will be given special attention.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-treatment stage as clinical IB-IIIA (AJCC/UICC 8th Edition);
2. Curative resectability has to be explicitly verified by the experienced surgical investigator;
3. Histologically confirmed diagnosis of primary non-small lung cancer.
4. Men and women aged 18 Years to 75 Years;
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1;
6. expected survival ≥ 6 months;
7. Sign on the informed consent form (ICF).

Exclusion Criteria:

1. Histologically confirmed were NOT NSCLC;
2. Lung cancer that can not be resected or has distant metastasis, or for other reasons can not tolerate surgery;
3. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colorectal, endometrial, cervical, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period;
4. Any active or history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications. The subjects were innate or acquired immunodeficiency (such as HIV), or active hepatitis (hepatitis B reference: HBsAg) positive; Hepatitis C reference: HCV antibody positive;
5. Uncontrolled diabetes or fasting blood glucose ≥11.0 mmol/L on the day of the test;
6. Women who are or may become pregnant, and lactating women are excluded;
7. Having a history of severe cardiovascular disease, severe myelosuppression and severe hepatic and renal insufficiency. Having a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
8. Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients requiring neoadjuvant immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | MPR will be assessed within 3 weeks after surgery
  Defined as the incidence rate in postoperative pathology where the percentage of surviving tumor cells in the tumor bed is ≤ 10%, regardless of the presence or absence of live tumor cells in the lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No